CLINICAL TRIAL: NCT07011797
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Phase 2 Study to Evaluate the Efficacy and Safety of CX11 Tablets in Overweight/Obese Participants
Brief Title: A Study to Evaluate the Efficacy and Safety of CX11 Tablets in Overweight/Obese Participants
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Corxel Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CX11201
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Obesity
Keywords: Overweight/Obese participants; Changes in weight and weight related indicators; Safety and Tolerability of IP; Efficacy, Safety, Tolerability and PK characteristic of different doses; Percentage change in weight; Body weight reduction; Change in waist circumference; Change in Body Mass Index; Pharmacokinetic analysis; Columbia-Suicide Severity Rating Scale; Patient Health Questionnaire-9; Weight loss
MeSH Terms: conditions — Obesity; Overweight; Weight Loss

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo group (Placebo Comparator)
  Interventions: Other: Placebo
- 120 mg group (Experimental)
  Interventions: Drug: CX11
- 160 mg group (Experimental)
  Interventions: Drug: CX11
- 200 mg fast titration group (Experimental)
  Interventions: Drug: CX11
- 200 mg slow titration group (Experimental)
  Interventions: Drug: CX11

INTERVENTIONS:
Drug: CX11 — CX11 tablets administered orally once daily (QD) with meals
  Other Names: VCT220
  Arms: 120 mg group; 160 mg group; 200 mg fast titration group; 200 mg slow titration group
Other: Placebo — Matching placebo tablets administered orally once daily (QD) with meals
  Arms: Placebo group

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled Phase 2 clinical study:

* To evaluate the efficacy of different dose levels of CX11 tablets in body weight reduction as compared to placebo.
* To compare the changes of effects in weight and weight-related indicators at the visit time points.
* To evaluate the tolerability and safety of different doses of CX11 tablets in overweight/obese participants.
* To assess the pharmacokinetics (PK) of different doses of CX11 tablets in overweight/obese participants.

Overweight/obese participants who are successfully screened will be randomized in a 1:1:1:1:1 ratio to different doses of CX11 tablets or placebo. All participants will enter a 2-week follow-up period after 36 weeks of treatment for safety observation.

ELIGIBILITY:
Inclusion Criteria

Participants who meet all of the following criteria will be eligible to participate in this study:

* Between 18 and 75 years old. Both men and women can participate, but women may make up to 70% of the participants.
* BMI of 30 or higher, or a BMI between 27 and 30 with at least one related health condition such as prediabetes, high blood pressure, abnormal cholesterol levels, fatty liver, or sleep apnea due to being overweight.
* HbA1c level below 6.5% and fasting blood sugar levels below 126 mg/dL.
* Have tried and failed to lose weight through diet and exercise at least once before the study and must have had a stable body weight (less than a 5% change) in the 90 days before the study.
* Participants and their partners must not plan to become pregnant or donate sperm/eggs during the study and for 90 days after. They must agree to use effective contraception for at least 6 months prior to screening and continue their chosen contraception method throughout the study. Women who could become pregnant must have a negative pregnancy test 24 hours before the first dose of study drug.
* Willing to maintain a stable diet and exercise routine during the study and keep a diary of their activities.
* Understand the study procedures, be willing to follow the study rules strictly, and sign a consent form voluntarily.

Exclusion Criteria

Participants who meet any of the following criteria will be excluded from this study:

* Known or suspected hypersensitivity to GLP-1 receptor agonists or similar products.
* Took part in another clinical study and received treatment within the last 90 days or within 5 drug elimination half-lives.
* Any type of diabetes.
* Obesity caused by hormonal or genetic issues such as thyroid problems, Cushing's syndrome, or other specific conditions.
* Have had or plan to have obesity treatment surgery or use weight loss devices, with some exceptions if done over a year ago.
* Have used certain medications or therapies for weight loss or conditions affecting weight, including GLP-1 receptor agonists and other related drugs, within the last 90 days.
* Recent serious heart problems, uncontrolled high blood pressure, or certain ECG abnormalities.
* History of pancreatitis, gallbladder disease (except for those treated with cholecystectomy), or evidence of hypothyroidism (except for participants who have normal thyroid function at screening and have been on a stable dose thyroid replacement for at least 90 days and are expected to maintain a stable dose during the study) or hyperthyroidism or thyrotoxicosis.
* History of cancer in the last 5 years, except for localized basal or squamous skin cancer, in situ carcinomas of the cervix, or in situ prostate cancer.
* Serious gastrointestinal diseases or surgeries that affect drug absorption.
* Active liver disease, excluding nonalcoholic fatty liver disease.
* Other serious health conditions that could increase study risk or make participation inappropriate, including certain psychiatric disorders.
* Recent history of unexplained fainting or family history of long QT syndrome or sudden death.
* History of organ transplant or severe autoimmune diseases.
* Had major surgery within the last 6 months or plan to have surgery soon.
* Significant abnormalities in kidney function, liver enzymes, blood tests, or other specified lab results.
* Positive for hepatitis B, hepatitis C, or HIV.
* Donated blood, lost a lot of blood, or received a transfusion in the last 90 days.
* Exceed weekly alcohol intake limits or have a history of drug abuse (including cannabis, its derivatives, or any cannabis-containing products; except for prescribed drug for medical purpose).
* Women who are pregnant or breastfeeding.
* Any other disease, condition, or medication that the investigator believes would interfere with the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2025-06-17 (Actual); Primary Completion 2026-03-23 (Estimated); Study Completion 2026-04-06 (Estimated)

PRIMARY OUTCOMES:
Percentage change in body weight from baseline | At Week 26

SECONDARY OUTCOMES:
Proportion of participants achieving ≥ 5% body weight reduction from baseline | At Week 26
Percentage change in body weight from baseline | At Week 36
Proportion of participants achieving ≥ 5% body weight reduction from baseline | At Week 36
Proportion of participants achieving ≥ 10% body weight reduction from baseline | At Week 26 and Week 36
Change in body weight from baseline | At Week 26 and Week 36
Change in waist circumference from baseline | At Week 26 and Week 36
Change in body mass index (BMI) from baseline | At Week 26 and Week 36
Number of adverse events (AEs) | Study duration, approximately 38 weeks
Number of treatment-emergent adverse events (TEAEs) | Study duration, approximately 38 weeks
Number of AE of special interest (AESI) | Study duration, approximately 38 weeks
Number of serious adverse events (SAEs) | Study duration, approximately 38 weeks
Columbia-Suicide Severity Rating Scale [C-SSRS] | At Day 1, Week 12, Week 26, Week 36 or at early termination (ET)
  Higher scores on the C-SSRS indicate a worse outcome, as they reflect greater severity of suicidal ideation and behavior. The scale begins at 0 and there is no single maximum value as the scale consists of multiple items that assess different aspects of suicidal ideation and behavior. Each item is scored individually, and the overall assessment is based on the combination of responses.
Patient Health Questionnaire-9 [PHQ-9] | At Day 1, Week 12, Week 26, Week 36 or at ET
  Higher scores on the PHQ-9 indicate a worse outcome, as they reflect more severe depression. The minimum score of the PHQ-9 is 0 and the maximum score of the PHQ-9 is 27.
Maximum steady-state plasma concentration (Cmax,ss) | Day 1 through Week 26
Minimum steady-state plasma concentration (Cmin,ss) | Day 1 through Week 26
Time to maximum steady-state plasma concentration (Tmax,ss) | Day 1 through Week 26
Area under the curve from 0 h to the time of the last quantifiable concentration (AUC0-last,ss) | Day 1 through Week 26
Area under the concentration-time curve over the dosing interval (AUC0-tau) | Day 1 through Week 26

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - AES - DRS - Synexus Clinical Research US, Inc. - Phoenix Central, Phoenix, Arizona
  - 310 Clinical Research - Alliance Clinical - Los Angeles, Inglewood, California
  - Acclaim Clinical Research - Alliance Clinical - San Diego, San Diego, California
  - Angels Clinical Research Institute - Miami, Doral, Florida
  - AES - DRS - Optimal Research Florida - Melbourne, Melbourne, Florida
  - Angels Clinical Research Institute, Miami, Florida
  - Palm Springs Community Health Center, Miami Lakes, Florida
  - Oceanic Research Group, LLC, North Miami Beach, Florida
  - Privia Medical Group Georgia, LLC - Savannah - Javara - PPDS, Savannah, Georgia
  - Privia Medical Group Georgia, LLC - Thomasville - Javara - PPDS, Thomasville, Georgia
  - Velocity Clinical Research - Valparaiso (Buynak Clinical Research) - PPDS, Valparaiso, Indiana
  - Mankato Clinic - East Main Street - Javara - PPDS, Mankato, Minnesota
  - Velocity Clinical Research - Cincinnati (Springdale) - Ohio - PPDS, Cincinnati, Ohio
  - Velocity Clinical Research - Dallas - PPDS, Dallas, Texas
  - Epic Clinical Research - Alliance Clinical - Lewisville, Lewisville, Texas
  - AES - DRS - Synexus Clinical Research US, Inc. - San Antonio, San Antonio, Texas
  - Flourish Research - San Antonio - PPDS, San Antonio, Texas